CLINICAL TRIAL: NCT04352751
Title: Experimental Use of Convalescent Plasma for Passive Immunization in Current COVID-19 Pandemic in Pakistan in 2020
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hilton Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PIPK- 0000 /NIBD-0000/2020
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-04

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Single arm, open label, clinical trial employing WHO recognized monitored emergency use of unregistered and experimental interventions (MEURI) study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Intervention: Convalescent plasma (Frozen Solution for infusion) obtained from COVID-19 recovered patients.
  The dosage depends upon the clinical situation and underlying disorder. Children: 15 ml/kg over 4-6 hours once in patients under 35 kg body weight. Adults: maximum 450 - 500 ml over 4-6 hours once in all adults patients.
  Interventions: Other: convalescent plasma

INTERVENTIONS:
Other: convalescent plasma — * Plasmapheresis, 900 - 1000 mL each time.
  * Standard apheresis plasma collection protocol using Haemonetics MCS+ intermittent blood flow system or Terumo Optia, Cobe-Spectra, Trima or Fresenius continuous flow system to be used.
  * Isovolumic saline replacement should be done.
  * Each donor can donate convalescent plasma again after an interval of every 2 weeks

SUMMARY:
Experimental Use of Convalescent Plasma of Passive Immunisation In Current COVID-19 Pandemic in Pakistan in 2020 Rationale & Objective: This study would help to gather real-life setting clinical data in local population, ultimately leading to increased evidence based management of the disease condition in the said population.

Eligibility:

1. informed consent must have been obtained
2. confirmed COVID-19 cases confirmed by RT-PCR laboratory tests
3. moderately severe or severe life-threatening COVID-19 related features: a) Moderately Severe disease as defined by the following features: i) Shortness of breath, ii) respiratory rate ≥ 30/min, iii) arterial blood oxygen saturation ≤ 92%, iv) and/or lung infiltrates > 25% within 24 to 48 hours 67 b) Severe Life-threatening disease as defined by: i) respiratory failure, ii) shock, and/or § multiple organ dysfunction

   Exclusion Criteria:

   Allergy history of plasma, sodium citrate and methylene blue; 2. For patients with history of autoimmune system diseases or selective IgA deficiency, 3. the application of convalescent plasma should be evaluated cautiously by clinicians.
4. Patients having evidence of uncontrolled cytokine release syndrome leading to end-stage multiorgan failure.

Methodology:

Total sample size is n=2000. A case report form (CRF) will have to be generated for each corona virus patient at baseline and the completion of study endpoint (at the time of discharge and at 4 weeks after experimental treatment modality using convalescent plasma.

* A unique identification number will be issued for each patient in this protocol.
* This data will be recorded in the national database. Data sources & Analysis: Patient data originating from patient medical record and assessments (mentioned in table below) will be recorded in the study CRF. Safety data (AEs and SAEs) from any time point during the study will be recorded in the study CRF. All analyses will be performed by third party statistician on SPSS. For continuous variables, summary statistics included n (number of observations), mean, standard deviation, median, minimum and maximum values, as well as frequencies and percentages for categorical variables will be presented.

DETAILED DESCRIPTION:
Passive immunization involves the administration of antibodies against a given agent to a susceptible individual for the purpose of preventing or treating an infectious disease due to that agent. A general principle of passive antibody therapy is that it is more effective when used for prophylaxis than for treatment of disease. When used for therapy, antibody is most effective when administered shortly after the onset of symptoms. The reason for temporal variation in efficacy is not well understood but could reflect that passive antibody works by neutralizing the initial inoculums, which is likely to be much smaller than that of established disease. As an example, passive antibody therapy for pneumococcal pneumonia was most effective when administered shortly after the onset of symptoms, and there was no benefit if antibody administration was delayed past the third day of disease.

The therapeutic benefits of convalescent plasma were formally studied in animal models in early 20th century. It efficacy was first determined in 1916, when 26 poliomyelitis patients were treated with convalescent plasma from polio survivors. Subsequently, therapeutic and prophylactic significance was explored in influenza and measles. Transfusion of immune plasma is a standard treatment modality for various viral hemorrhagic fevers. Its efficacy in treating Ebola Virus Disease is also well established. Studies have reported reduction viral load in patients with H1N1 influenza. Of special attention is the meta-analysis, carried out by Mair-Jenkinset al, concluding effectiveness of passive immunization as a treatment option for severe viral acute respiratory infections caused by SARS corona virus, influenza A (H1N1), avian influenza A (H5N1) and Spanish influenza A. Efficacy of convalescent plasma has been anecdotally reported in SARS-CoV-2 infections.

ELIGIBILITY:
Inclusion Criteria:

FOR DONORS:

1. Volunteer enrolment (Informed consent will be obtained; Annexures-2A & 2B).
2. All the regulations related to ICH-GCP and Blood Transfusion Authority (BTA) Pakistan will be followed.
3. Should fulfill all the criteria of a healthy blood donor (with the exception of history of COVID-19 during last 4-8 weeks.
4. History of COVID-19 during last 4-8 weeks
5. RT-PCR negative for SARS-CoV-2 RNA (carried out on nasopharyngeal or oropharyngeal specimen)
6. Age cutoff: 18-55years
7. Body weight cut off: >50 kg for men and > 45kg for women

FOR RECIPIENTS:

1. Volunteer enrolment (Informed consent will be obtained; Annexures-3A & 3B).
2. Confirmed COVID-19 cases confirmed by RT-PCR laboratory tests
3. Severe or Critical COVID-19 related features (8):

   a. Severe COVID-19, defined by the presence of any of the following features: i. Shortness of breath ii. Respiratory rate ≥ 30/min, iii. Arterial blood oxygen saturation ≤ 93%, iv. Lung infiltrates > 50% within 24 to 48 hours b. CriticalCOVID-19, defined by the presence of any of the following features: i. Respiratory failure, ii. Shock iii. Multiple organ dysfunction

Exclusion Criteria:

1. Allergy history for plasma, sodium citrate and methylene blue
2. For patients with history of autoimmune system diseases or selective IgA deficiency, the application of convalescent plasma should be evaluated cautiously by clinicians.
3. Patients having evidence of uncontrolled cytokine release syndrome leading to end-stage multi organ failure.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2000 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Change in COVID-19 severity status | Up to 09 days
  Improvement in disease severity will be regarded as a shift from Critical to Severe or from Severe to Mild disease category. The various disease categories are defined as following (17):
  1. Mild COVID-19, defined by the absence of features given in criteria for moderate and severe disease.
  2. Severe COVID-19, defined by the presence of any of the following features:
  i. Shortness of breath ii. Respiratory rate ≥ 30/min, iii. Arterial blood oxygen saturation ≤ 93%, iiii. Lung infiltrates > 50% within 24 to 48 hours c. Critical COVID-19, defined by the presence of any of the following features: i. Respiratory failure, ii. Shock iii. Multiple organ dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tahir Shamsi, FRCP MRCPath, Principal Investigator — National Institute of Blood Diseases and Bone Marrow Transplantation (NIBD)
Locations (1):
- National Institute of Blood Diseases and Bone Marrow Transplantation (NIBD), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robbins JB, Schneerson R, Szu SC. Perspective: hypothesis: serum IgG antibody is sufficient to confer protection against infectious diseases by inactivating the inoculum. J Infect Dis. 1995 Jun;171(6):1387-98. doi: 10.1093/infdis/171.6.1387. PMID 7769272
- [Background] Casadevall A, Scharff MD. Serum therapy revisited: animal models of infection and development of passive antibody therapy. Antimicrob Agents Chemother. 1994 Aug;38(8):1695-702. doi: 10.1128/AAC.38.8.1695. No abstract available. PMID 7985997
- [Background] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066
- [Background] Luke TC, Casadevall A, Watowich SJ, Hoffman SL, Beigel JH, Burgess TH. Hark back: passive immunotherapy for influenza and other serious infections. Crit Care Med. 2010 Apr;38(4 Suppl):e66-73. doi: 10.1097/CCM.0b013e3181d44c1e. PMID 20154602
- [Derived] Khan TNS, Mukry SN, Masood S, Meraj L, Devrajani BR, Akram J, Fatima N, Maqsood S, Mahesar A, Siddiqui R, Ishaque S, Afzal MB, Mukhtar S, Ahmed S, Naz A, Shamsi TS. Usefulness of convalescent plasma transfusion for the treatment of severely ill COVID-19 patients in Pakistan. BMC Infect Dis. 2021 Sep 27;21(1):1014. doi: 10.1186/s12879-021-06451-7. PMID 34579646